CLINICAL TRIAL: NCT04509479
Title: National Tunisian Registry of Valvulopathies (NATURE-VALVE)
Acronym: NATURE-VALVE
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society of Cardiology and Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: DAC-008-STCCCV
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Valvular Heart Disease; Valvular Stenosis; Valvular Insufficiency
Keywords: Valvular; Heart; Aortic; Mitral; Tricuspid
MeSH Terms: conditions — Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Valve replacement — Description of valve replacements

SUMMARY:
The National Tunisian Registry of Valvulopathies is an observational, prospective and multicenter study aiming to assess the epidemiological, clinical and therapeutic profile of valve disease in tunisian departments of cardiology. Cardiologists from both sectors (public and private) are participating in the study, with 37 investigational centers. Data will be captured electronically by DACIMA Clinical Suite, according to FDA 21 CFR part 11 (Food and Drug Administration 21 Code of Federal Regulations part 11), HIPAA (Health Insurance Portability and Accountability Act) & ICH (International Conference on Harmonisation) requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients originated from Tunisia
* Signed informed consent
* Patients with at least one of the following conditions :

  1. moderate to severe native mitral and / or aortic and / or tricuspid native valve disease
  2. and / or a history of a previous percutaneous or surgical valve intervention
  3. and / or a history of infectious endocarditis

Exclusion Criteria:

* Congenital valve diseases not including bicuspid aortic valve
* Isolated pulmonary valvulopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with valvular disease
Sampling Method: Non-Probability Sample
Enrollment: 3637 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Valvulopathies incidence | at inclusion
  Number of subjects with valvular disease (mitral or aortic or tricuspid) and willing to participate at the study

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | at 6 months of follow-up
  Number of patients with Major adverse cardiovascular events (MACE), including nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death.

CONTACTS AND LOCATIONS:
Overall Officials: Fathia Mghaieth, MD, Study Chair — Tunisian Society of Cardiology and Cardiovascular Surgery; Lilia Zakhama, MD, Study Chair — Tunisian Society of Cardiology and Cardiovascular Surgery
Locations (1):
- The Tunisian Society of Cardiology and CardioVascular Surgery, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No